CLINICAL TRIAL: NCT02788110
Title: Prospective Crossover Comparison of Work of Breathing During Non-invasive Ventilation: Neurally Adjusted Ventilatory Assist (NAVA) Versus Nasal Intermittent Positive Pressure Ventilation (NIPPV) in Premature Neonates
Brief Title: Work of Breathing During Non-invasive Ventilation in Premature Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB 205507
Record Dates: First submitted 2016-05-23; First posted 2016-06-02 (Estimated); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Respiratory Distress Syndrome, Newborn; Bronchopulmonary Dysplasia
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn; Bronchopulmonary Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NIV NAVA then NIPPV (Other): Infants will receive 15 minute trials of noninvasive neurally adjusted ventilatory assist (NIV NAVA) and nasal intermittent positive pressure ventilation (NIPPV) in random order with the first 10 minutes after changing to be considered a washout period and the last 5 minutes used for data collection. This group will receive NIV NAVA then NIPPV.
  Interventions: Other: Noninvasive neurally adjusted ventilatory assist (NIV NAVA); Other: Nasal intermittent positive pressure ventilation (NIPPV)
- NIPPV then NIV NAVA (Other): Infants will receive 15 minute trials of noninvasive neurally adjusted ventilatory assist (NIV NAVA) and nasal intermittent positive pressure ventilation (NIPPV) in random order with the first 10 minutes after changing to be considered a washout period and the last 5 minutes used for data collection. This group will receive NIPPV then NIV NAVA.
  Interventions: Other: Noninvasive neurally adjusted ventilatory assist (NIV NAVA); Other: Nasal intermittent positive pressure ventilation (NIPPV)

INTERVENTIONS:
Other: Noninvasive neurally adjusted ventilatory assist (NIV NAVA) — Neurally adjusted ventilatory assist (NAVA) is a mode of ventilation that uses a functional naso/orogastric tube with embedded electrodes which detect diaphragmatic contractions (called the Edi signal). NAVA uses this Edi signal to synchronize ventilator support to the patient's own respiratory efforts and to support these efforts as needed.
Other: Nasal intermittent positive pressure ventilation (NIPPV) — Nasal intermittent positive pressure ventilation (NIPPV) or noninvasive pressure control ventilation (NIV PC) is a mode of ventilation delivering unsynchronized puffs of air or "breaths" to a baby through nasal cannulae.
  Other Names: Noninvasive pressure control ventilation (NIV PC)

SUMMARY:
Background:

Non-invasive forms of respiratory support have been developed to manage respiratory distress and failure in premature newborns without exposing them to the risks associated with invasive mechanical ventilation. It has been difficult to synchronize non-invasive ventilation due to the large air leaks, high respiratory rates, and small tidal volumes inherent to this interface and population. Neurally adjusted ventilatory assist (NAVA) is a novel mode of ventilation that uses a functional naso/orogastric tube with embedded electrodes which detect diaphragmatic contractions (called the Edi signal). NAVA uses this Edi signal to synchronize ventilator support to the patient's own respiratory efforts and to support these efforts as needed. Few studies have examined the use of NAVA with non-invasive ventilation (NIV) in preterm neonates. A group at Arkansas Children's Hospital recently completed a study, looking at work of breathing in an animal model comparing NIV NAVA with the unsynchronized nasal intermittent positive pressure (NIPPV) mode currently used at this hospital. They were able to show that work of breathing was lower with NAVA in this model. This study will take what was shown in the animal model and translate this to the bedside. Using respiratory inductance plethysmography to measure thoracoabdominal asynchrony, this study will compare work of breathing during NIPPV versus NIV NAVA in preterm neonates with respiratory insufficiency.

Hypothesis:

Work of breathing as estimated by the phase angle (θ) using respiratory inductance plethysmography will be decreased with the use of NIV NAVA in comparison to unsynchronized NIPPV in premature neonates with respiratory insufficiency.

Methods:

Fifteen premature neonates of between 1-2 kilograms' current weight, with gestational age at birth between 24-34 weeks, and receiving non-invasive ventilation will be enrolled in the study after consent is obtained. The infants will be ventilated using NIV NAVA and NIPPV applied in random order for 15 minutes each while using respiratory inductance plethysmography to measure thoracoabdominal asynchrony as an estimate of work of breathing.

Significance:

This study will identify whether or not NIV NAVA has advantages over NIPPV for improving work of breathing in premature neonates.

DETAILED DESCRIPTION:
Background/Rationale:

Historically, respiratory insufficiency and respiratory failure have been frequent sources of morbidity and mortality in premature neonates. Intubation for invasive mechanical ventilation has been a life-saving therapy for many of these patients, but is not without risks. These risks include pulmonary complications such as volutrauma, extrapulmonary air leak syndromes, and traumatic injury to the large airways; non-pulmonary complications such as retinopathy of prematurity; and long-term complications such as bronchopulmonary dysplasia [Miller, Badiee]. Concern over these effects of prolonged mechanical ventilation has led to the development of non-invasive forms of respiratory support.

Non-invasive ventilation (NIV) is a frequently used modality of respiratory support for premature neonates in the setting of respiratory insufficiency or recent weaning from invasive ventilation. Synchronized NIV is effective at decreasing respiratory effort as compared to unsynchronized NIV and nasal continuous positive airway pressure (NCPAP) [Chang]. Synchronizing NIV in premature neonates to the patient's own respiratory efforts is difficult because of the large air leaks, weak inspiratory efforts, and high respiratory rates inherent to this population [Vignaux].

A novel method of synchronization, neurally adjusted ventilatory assist (NAVA) uses electrodes on a functional naso/orogastric tube (Edi catheter) to detect diaphragm contractions and time the onset, duration, and peak inspiratory pressure of supporting breaths with the electrical activity of the diaphragm (Edi) [Sinderby]. NAVA can be used with both invasive and non-invasive ventilation modalities, and there have been several small studies examining invasive NAVA in children and adults [Stein, de la Olivia]. Fewer studies have examined NIV NAVA in these populations, and only two clinical trials have examined NIV NAVA in premature neonates [Beck, Lee]. Beck and colleagues in Canada showed feasibility and preservation of synchrony during NIV NAVA in premature neonates [Beck]. Lee and colleagues in Korea showed fewer asynchrony events, lower trigger delay, and lower peak inspiratory pressures with NIV NAVA compared to non-invasive pressure support ventilation in premature neonates [Lee]. Neither study examined work of breathing (WOB) in preterm neonates ventilated with NIV NAVA.

Work of breathing during assisted ventilation is the portion of the driving pressure for ventilation contributed by the patient's respiratory muscles. A research team at Arkansas Children's Hospital was able to demonstrate that NAVA achieves reduced response time, work of breathing, and asynchrony with neurally triggered breaths as compared to pneumatically triggered breaths in an animal model [Heulitt]. This team was also able to show similar results in a clinical study of intubated pediatric patients with bronchiolitis [Clement]. A recently completed study at this institution looked at work of breathing in neonatal pigs comparing NIV NAVA with the unsynchronized nasal intermittent positive pressure (NIPPV) mode currently used at this hospital. Using the pressure-time product (PTP) as a measure of WOB this study was able to show that WOB was lower with NAVA. The PTP cannot be reliably used in infants on NIV because the nasal prong interface allows large air leaks at the nose and mouth, which interfere with accurate measurements.

Thoracoabdominal asynchrony (TAA) is an important correlate of WOB and increased respiratory load in preterm infants and can be measured without invasive monitoring. TAA can be measured using a respiratory inductance plethysmography (RIP) bands around the patient's chest and abdomen to quantify chest wall and abdominal movement. The degree of asynchrony between the two compartments is reflected in the phase angle (θ), which can be calculated from the RIP band measurements.

This study will examine estimated WOB in a population of premature neonates with respiratory insufficiency currently on non-invasive support. Infants will serve as their own controls and will be studied on NIV NAVA and NIPPV. Order of assignment will be randomized. Researchers will use RIP bands to measure thoracic and abdominal movement, then calculate the phase angle (θ) as an estimate of WOB. Study personnel will measure other respiratory parameters correlating with ventilation and gas exchange including the following: tidal volume (arbitrary units, AU), minute ventilation (AU/min), respiratory rate, transcutaneous oxygen and carbon dioxide, oxygen saturation and FiO2 requirement, peak inspiratory pressure, and delivered end expiratory pressure. Investigators will also evaluate measures of breathing asynchrony to include trigger delay (time between initial increase in Edi signal and initiation of delivered ventilator flow) and asynchrony index (number of asynchrony events divided by total events, as a percent).

Study Design/Procedures/Population:

Fifteen premature neonates of between 1-2 kilogram current weight, with gestational age at birth between 24-34 weeks, and receiving non-invasive ventilation will be enrolled in the study. Inclusion criteria will be as follows: respiratory insufficiency currently requiring non-invasive ventilation (either NIPPV or NAVA), current FiO2 requirement less than 0.40, and clinical stability. Exclusion criteria will be as follows: ionotropic support, clinical instability (temperature instability, heart failure, bleeding, active infection, significant apnea or bradycardia), known major congenital anomalies (congenital heart disease, abdominal wall defects, gastrointestinal tract defects, cleft palate, or neurologic defects), known cystic fibrosis, nitric oxide use, and cyanotic congenital heart disease.

At the beginning of the study, RIP bands will be placed around the infant's chest and abdomen. An Edi catheter will be placed and the current gastric catheter may or may not be removed. Infants will be ventilated with the Servo i ventilator equipped with NIV NAVA software {Maquet, Solna, Sweden}. Data will be continuously and simultaneously acquired using the MP100 Biopac data acquisition system. Data acquired will be as follows: heart rate, oxygen saturation, transcutaneous CO2 and O2, PIP, PEEP, rib cage and abdominal RIP signals, summed tidal volume, and Edi. Infants will receive 15 minute trials of NIV NAVA and NIPPV in random order with the first 10 minutes after changing to be considered a washout period and the last 5 minutes used for data collection. The data recorded from the two RIP bands will be used to calculate the phase angle (θ) as an estimate of WOB.

Risks and Benefits:

Infants often have gagging and may have vomiting when a gastric tube, such as the NAVA catheter, is removed or replaced. Rarely, patients could have a gastric tube go into a place besides the stomach or coil in the esophagus. Researchers should be able to detect if this occurs using the placement screen on the ventilator because the NAVA catheter has electrodes on it that detect the electrical activity of the heart and diaphragm, which can be used to determine the location.

In extremely low birth weight infants, transcutaneous monitors (TCOMs) can cause skin burning. These effects are not seen in larger babies like those included in this study.

There is a small risk of loss of confidentiality inherent in all research. Investigators will do everything possible to protect the participants' confidentiality.

There may or may not be direct medical benefit to the infants involved in this study. The infants will have continuous carbon dioxide and oxygen monitoring during the study and if any patient has any problems, study personnel will be able to detect and respond to this quickly. If a patient shows improvement while using NAVA, investigators may be able to suggest to the treatment team that this mode be continued. If using NAVA improves work of breathing in babies, then the researchers hope the information learned from this study will benefit other infants needing respiratory support in the future.

Data Handling/Recordkeeping:

The principal investigator will carefully monitor study procedures to protect the safety of research subjects, the quality of the data and the integrity of the study. Each patient will be assigned a unique identifying code or number. The key to the code will be kept in a locked file in the principal investigator's office. Only the principal investigator and co-investigators will have access to the code and information that identifies the subject in the study.

Data Analysis:

The primary hypothesis is that phase angle (θ) using respiratory inductance plethysmography will be decreased with the use of NAVA in comparison to NIPPV in our study sample.

Data collected will be checked for outliers and extreme values, as well as distributional assumptions of the parametric statistical tests. Repeated measures ANOVA will be used to compare the primary and secondary outcomes under the two ventilation methods when such assumptions are met. When significant deviation from assumptions is encountered, nonparametric alternatives will be used. Statistical analyses will be performed using Stata (College Station, TX) statistical software.

Sample Size, Power Calculation:

Investigators plan to recruit 15-20 neonates who are 24-34 weeks gestation with respiratory insufficiency. Based on the results in the animal model, a 30% reduction in the primary outcome is expected. Since the average phase angle was found to be variable among preterm infants (ranged from 2.8-162.9), there are several scenarios of the sample size and power calculation presented for analysis [Ulm]. A sample size of 15 neonates achieves 82% power to detect a 30% change in the primary outcome with an estimated standard deviation of differences of 18.8, 37.5, or 56.3 respectively for an average phase angle of 50, 100, and 150 degrees with the use of NIPPV. All calculations assume a significance level of 0.05 using a two-sided paired t-test.

Ethical Considerations:

This study will be conducted in accordance with all applicable government regulations and University of Arkansas for Medical Sciences (UAMS) research policies and procedures. This protocol and any amendments will be submitted and approved by the UAMS Institutional Review Board (IRB). The formal consent of each subject, using the IRB-approved consent form, will be obtained before that subject is submitted to any study procedure. All subjects for this study will be provided a consent form describing this study and providing sufficient information in language suitable for subjects to make an informed decision about their participation in this study. The person obtaining consent will thoroughly explain each element of the document and outline the risks and benefits, alternate treatment(s), and requirements of the study. The consent process will take place in a quiet and private room or by phone, and subjects may take as much time as needed to make a decision about their participation. Phone consent will be obtained with a witness and consent will be faxed to parent(s). Phone consent will only be obtained in the event that the parents are unable to be present.

Participation privacy will be maintained and questions regarding participation will be answered. No coercion or undue influence will be used in the consent process. The consent form must be signed by the subject, the parent and the individual obtaining the consent. A copy of the signed consent will be given to the participant, and the informed consent process will be documented in each subject's research record.

Dissemination of Data:

Results of this study may be used for presentations, posters, or publications. The publications will not contain any identifiable information that could be linked to a participant.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age at birth between 24 and 34 weeks
* Receiving noninvasive ventilation
* Between 1 and 2 kg current weight
* Current FiO2 requirement less than 0.40
* Clinical stability

Exclusion Criteria:

* Known major congenital anomalies (congenital heart disease, abdominal wall defects, gastrointestinal tract defects, cleft palate, or neurologic defects)
* Clinical instability (temperature instability, heart failure, bleeding, active infection, significant apnea or bradycardia)
* Known cystic fibrosis
* Use of inhaled nitric oxide
* Cyanotic congenital heart disease

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Phase angle (θ) | 30 minutes
  The primary outcome of interest is phase angle (θ). Phase angle is reflective of work of breathing. Respiratory inductance plethysmography (RIP) signals will be analyzed as sine waves of the same frequency for the phase angle as follows: θ = (δt/P) x 360 degrees, where δt represents the time shift between the two sine waves and P is the wave period or cycle time.

SECONDARY OUTCOMES:
Tidal volume (arbitrary units, AU) | 30 minutes
  Tidal volume (arbitrary units, AU) measured by respiratory inductance plethysmography
Minute ventilation (AU/min) | 30 minutes
  Minute ventilation (AU/min) measured by respiratory inductance plethysmography
Respiratory rate (breaths/min) | 30 minutes
  Respiratory rate (breaths/min)
Transcutaneous oxygen (mmHg) | 30 minutes
  Transcutaneous oxygen (mmHg)
Transcutaneous carbon dioxide (mmHg) | 30 minutes
  Transcutaneous carbon dioxide (mmHg)
Oxygen saturation (%) | 30 minutes
  Oxygen saturation (%) measured by pulse oximetry
Peak inspiratory pressure (cmH2O) | 30 minutes
  Peak inspiratory pressure (cmH2O)
Positive end expiratory pressure (cmH2O) | 30 minutes
  Positive end expiratory pressure (cmH2O)
Trigger delay (ms) | 30 minutes
  Trigger delay (ms)
Asynchrony index (%) | 30 minutes
  Total number of asynchrony events divided by sum of ventilator cycles and ineffective efforts expressed as a percentage

CONTACTS AND LOCATIONS:
Overall Officials: David N Matlock, MD, Principal Investigator — University of Arkansas
Locations (1):
- Arkansas Children's Hospital, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miller JD, Carlo WA. Pulmonary complications of mechanical ventilation in neonates. Clin Perinatol. 2008 Mar;35(1):273-81, x-xi. doi: 10.1016/j.clp.2007.11.004. PMID 18280886
- [Background] Badiee Z, Nekooie B, Mohammadizadeh M. Noninvasive positive pressure ventilation or conventional mechanical ventilation for neonatal continuous positive airway pressure failure. Int J Prev Med. 2014 Aug;5(8):1045-53. PMID 25489454
- [Background] Chang HY, Claure N, D'ugard C, Torres J, Nwajei P, Bancalari E. Effects of synchronization during nasal ventilation in clinically stable preterm infants. Pediatr Res. 2011 Jan;69(1):84-9. doi: 10.1203/PDR.0b013e3181ff6770. PMID 20924313
- [Background] Vignaux L, Grazioli S, Piquilloud L, Bochaton N, Karam O, Levy-Jamet Y, Jaecklin T, Tourneux P, Jolliet P, Rimensberger PC. Patient-ventilator asynchrony during noninvasive pressure support ventilation and neurally adjusted ventilatory assist in infants and children. Pediatr Crit Care Med. 2013 Oct;14(8):e357-64. doi: 10.1097/PCC.0b013e3182917922. PMID 23863816
- [Background] Sinderby C, Beck J. Neurally adjusted ventilatory assist in non-invasive ventilation. Minerva Anestesiol. 2013 Aug;79(8):915-25. Epub 2013 Apr 5. PMID 23558763
- [Background] Stein H, Alosh H, Ethington P, White DB. Prospective crossover comparison between NAVA and pressure control ventilation in premature neonates less than 1500 grams. J Perinatol. 2013 Jun;33(6):452-6. doi: 10.1038/jp.2012.136. Epub 2012 Oct 25. PMID 23100042
- [Background] de la Oliva P, Schuffelmann C, Gomez-Zamora A, Villar J, Kacmarek RM. Asynchrony, neural drive, ventilatory variability and COMFORT: NAVA versus pressure support in pediatric patients. A non-randomized cross-over trial. Intensive Care Med. 2012 May;38(5):838-46. doi: 10.1007/s00134-012-2535-y. Epub 2012 Apr 6. PMID 22481227
- [Background] Beck J, Reilly M, Grasselli G, Mirabella L, Slutsky AS, Dunn MS, Sinderby C. Patient-ventilator interaction during neurally adjusted ventilatory assist in low birth weight infants. Pediatr Res. 2009 Jun;65(6):663-8. doi: 10.1203/PDR.0b013e31819e72ab. PMID 19218884
- [Background] Lee J, Kim HS, Jung YH, Shin SH, Choi CW, Kim EK, Kim BI, Choi JH. Non-invasive neurally adjusted ventilatory assist in preterm infants: a randomised phase II crossover trial. Arch Dis Child Fetal Neonatal Ed. 2015 Nov;100(6):F507-13. doi: 10.1136/archdischild-2014-308057. Epub 2015 Jul 15. PMID 26178463
- [Background] Heulitt MJ, Clement KC, Holt SJ, Thurman TL, Jo CH. Neurally triggered breaths have reduced response time, work of breathing, and asynchrony compared with pneumatically triggered breaths in a recovering animal model of lung injury. Pediatr Crit Care Med. 2012 May;13(3):e195-203. doi: 10.1097/PCC.0b013e318238b40d. PMID 22079957
- [Background] Clement KC, Thurman TL, Holt SJ, Heulitt MJ. Neurally triggered breaths reduce trigger delay and improve ventilator response times in ventilated infants with bronchiolitis. Intensive Care Med. 2011 Nov;37(11):1826-32. doi: 10.1007/s00134-011-2352-8. Epub 2011 Sep 23. PMID 21946913
- [Background] Ulm LN, Hamvas A, Ferkol TW, Rodriguez OM, Cleveland CM, Linneman LA, Hoffmann JA, Sicard-Su MJ, Kemp JS. Sources of methodological variability in phase angles from respiratory inductance plethysmography in preterm infants. Ann Am Thorac Soc. 2014 Jun;11(5):753-60. doi: 10.1513/AnnalsATS.201310-363OC. PMID 24716708
- [Derived] Matlock DN, Bai S, Weisner MD, Comtois N, Beck J, Sinderby C, Courtney SE. Work of Breathing in Premature Neonates: Noninvasive Neurally-Adjusted Ventilatory Assist versus Noninvasive Ventilation. Respir Care. 2020 Jul;65(7):946-953. doi: 10.4187/respcare.07257. Epub 2020 Feb 18. PMID 32071130